CLINICAL TRIAL: NCT05344391
Title: Can BFR Training on a Bike Augment RC Strength, Leg Strength, and VO2 Peak
Brief Title: BFR Training on a Bike to Augment RC Strength, Leg Strength, and VO2 Peak
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Jason Brumitt, Associate Professor of Physical Therapy, George Fox University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: George Fox College of PT
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Can BFR Cycling Augment Strength and VO2peak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR cycling (Experimental): This group will perform cycling with BFR applied bilaterally at 80% LOP for 10 min and cycling at 40% HRR. Next they will perform 3x15 of the scaption and sidelying external rotation exercises. These will initially be performed at 30% 1RM; every 2 weeks load increased by 1lbs.
  Interventions: Other: BFR cycling
- Cycling without BFR (Active Comparator): This group will perform cycling and the same shoulder exercises using the same training parameters; however, BFR will not be applied.
  Interventions: Other: Cycling without BFR

INTERVENTIONS:
Other: BFR cycling — Cycling with BFR followed by shoulder exercises
  Arms: BFR cycling
Other: Cycling without BFR — Cycling without BFR followed by shoulder exercises
  Arms: Cycling without BFR

SUMMARY:
This study will investigate if subjects who bike at 40% of heart rate reserve (HRR) with blood flow restriction (BFR) applied to bilateral thighs for 10 minutes (at 80% limb occlusion pressure) will experience greater gains in 10 rep max for dominant lower extremity leg press, greater gains in rotator cuff strength (hand held dynamometer testing for supraspinatus and external rotators) and greater gains in VO2 peak.

DETAILED DESCRIPTION:
This study will randomize healthy adult subjects to one of two groups: a BFR biking group that performs 10 min of cycling at 40% heart rate reserve (HRR) with bilateral occlusion applied to the proximal thighs (80% LOP) or to a non-biking BFR group perform 10 min of cycling at 40% HRR. After each cycling session subjects will perform 3x15 of the scaption exercise and 3x15 sidelying external rotation with their dominant upper extremity. They will initially start training the shoulder at 30% of 1RM (estimated from an equation formula) for the first 2 weeks followed by increasing training load by 1lbs each exercise every 2 weeks. The training program will last 6 weeks (3x week for 6 weeks, total of 18 sessions).

Pretest and posttests will include: VO2 peak testing on a cycle using Cosmed metabolic cart, hand held dynamometry to measure strength of the supraspinatus and external rotators of the shoulder using traditional manual muscle test positions, and on a separate day 10RM testing on a leg press for the dominant lower extremity.

ELIGIBILITY:
Inclusion Criteria: healthy adults (18 yrs of age and older) -

Exclusion Criteria: no current musculoskeletal symptoms/injuries; no prior lower extremity or shoulder/upper extremity surgery (dominant) during the prior year; no contraindications to BFR training

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
VO2peak | 6 weeks
  Pretest/posttest measures of VO2peak performance on the bicycle using Cosmed Metabolic Cart
Shoulder Strength | 6 weeks
  Using a Hand Held Dynamometer; shoulder strength will be measured pretest/posttest for teh supraspinatus and the shoulder external rotators (dominant UE)
10 RM unilateral leg press for the dominant lower extremity | 6 weeks
  Test 10 RM strength on the leg press for the dominant LE/ pretest/posttest

CONTACTS AND LOCATIONS:
Overall Officials: JASON BRUMITT, PhD, Principal Investigator — George Fox University
Locations (2):
- United States (2):
  - College of Physical Therapy / George Fox University, Newberg, Oregon
  - George Fox University School of Physical Therapy, Newberg, Oregon

IPD SHARING:
Plan to Share IPD: No